CLINICAL TRIAL: NCT03475758
Title: Phase II Study of Goserelin for Ovarian Protection in Premenopausal Patients Receiving Cyclophosphamide Containing Chemotherapy: Menstruation Outcome
Brief Title: Goserelin for Ovarian Protection in Premenopausal Patients Receiving Cyclophosphamide
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ashraf Saadeldin, assisstant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GOP
Record Dates: First submitted 2018-03-11; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Ovarian Failure
MeSH Terms: interventions — Goserelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chemotherapy without goserelin (No Intervention): these patients will receive their chemotherapy without addition of Goserelin
- chemotherapy with goserelin (Experimental): these patients will receive their chemotherapy with addition of Goserelin
  Interventions: Drug: Goserelin

INTERVENTIONS:
Drug: Goserelin — adding goserelin with chemotherapy
  Other Names: zoladex
  Arms: chemotherapy with goserelin

SUMMARY:
The use of adjuvant chemotherapy in younger women with early breast cancer (EBC) has substantially improved the long-term outcome. However, this benefit is associated with long-term toxic effects which are becoming more important as prognosis improves. These include premature menopause and infertility in young pre-menopausal women. The incidence of premature menopause depends on the type and intensity of chemotherapy and the patient's age. In women <35 years old, the long-term (3 years after diagnosis) incidence of amenorrhea is similar to women who have not received chemotherapy, at ∼ 10%, but this increases to 50% in women between 35 and 40 years old, and can be up to 85% in women >40 years. Premature ovarian failure has major consequences including sexual dysfunction and infertility, and the latter may be of great concern to younger patients with breast cancer and has a bearing in influencing treatment decisions in almost 30% of cases.

Currently, there is no standard treatment for preventing chemotherapy-induced ovarian failure. Previous studies have suggested that temporary ovarian suppression with a gonadotropin-releasing hormone (GnRH) analogue may preserve ovarian function both in humans and animal models. Clinical data are conflicting. For example, a recent Italian multi-center phase III study Prevention of Menopause-Induced by Chemotherapy: A Study in Early Breast Cancer Patients-Gruppo Italiano Mamella 6 (PROMISE-GIM6) reported that the use of GnRH analogue, triptorelin during chemotherapy in pre-menopausal patients with EBC, reduced the occurrence of chemotherapy-induced early menopause with four pregnancies after a 26-month follow-up [one in the chemotherapy alone arm and three in the triptorelin with chemotherapy arm]. In contrast, another trial suggested that the use of goserelin concurrently with neoadjuvant chemotherapy did not significantly reduce incidence of amenorrhea 6 months after the end of chemotherapy compared with those receiving chemotherapy alone and only two pregnancies were recorded [one in each arm] with a follow-up of 2 years.

DETAILED DESCRIPTION:
In this phase II trial, patients will be randomly assigned, in a 1:1 ratio, to standard adjuvant or neoadjuvant chemotherapy with the GnRH agonist goserelin (goserelin group) or to chemotherapy without goserelin (chemotherapy alone group).

For Patients randomly assigned to the goserelin group, goserelin at a dose of 3.6 mg will be administered subcutaneously every 4 weeks beginning 1 week before the initial chemotherapy dose and will be continued to within 2 weeks before or after the final chemotherapy dose.

Follow up: All patients will be followed for at least 1 year clinically monthly and by laboratory assessment by hormonal profile (FSH, LH, E2) every 6 months.

ELIGIBILITY:
Inclusion Criteria:

Premenopausal cancer patients who will receive Cyclophosphamide-containing chemotherapy.

Exclusion Criteria:

postmenopausal cancer patients. cancer patients who will receive non Cyclophosphamide containing chemotherapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — premenopausal patients
Enrollment: 100 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
compare rate of ovarian failure at 1 year between the two treatment groups | 1 year
  rate of ovarian failure

CONTACTS AND LOCATIONS:
Overall Officials: samir Eid, phd, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Peto R, Davies C, Godwin J, Gray R, Pan HC, Clarke M, Cutter D, Darby S, McGale P, Taylor C, Wang YC, Bergh J, Di Leo A, Albain K, Swain S, Piccart M, Pritchard K. Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100,000 women in 123 randomised trials. Lancet. 2012 Feb 4;379(9814):432-44. doi: 10.1016/S0140-6736(11)61625-5. Epub 2011 Dec 5. PMID 22152853

DOCUMENTS (1):
  • Study Protocol (2018-03-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT03475758/Prot_000.pdf